CLINICAL TRIAL: NCT00183001
Title: Effect of Vitamin K on Age-Related Bone Loss and Vascular Calcification
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Arthritis Foundation (Other); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0048; R01AG019147 (NIH); R01HL069272 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Osteoporosis; Vascular Calcification; Inflammation
Keywords: nutritional supplement; dietary supplement; vitamin therapy; Vitamin K deficiency; bone density
MeSH Terms: conditions — Osteoporosis; Vascular Calcification; Inflammation; Vitamin K Deficiency | interventions — Vitamin K

INTERVENTIONS:
Drug: Vitamin K

SUMMARY:
The purpose of this study is to determine if supplemental vitamin K will reduce age-related bone loss in elderly men and women above that achieved by supplementation.

DETAILED DESCRIPTION:
This is a three-year, double-blind, placebo-controlled trial to study the effect of vitamin K supplementation (500 µg/d) on bone density at the hip, markers of bone turnover, vascular calcification, osteoarthritis and tests of concentration in 452 men and women, aged 60-80 years. All participants will also be receiving calcium and vitamin D supplements, in addition to a multivitamin, to prevent any potential bone loss associated with dietary inadequacy of these nutrients.

Measurements of plasma vitamin K concentrations, percent undercarboxylated osteocalcin (markers of vitamin K status), serum osteocalcin, collagen Type-I-crosslink N-telopeptides (markers of bone turnover) and BMD of the hip, as well as the heel, spine and total body at 0, 6, 12, 24, and 36 months of vitamin K supplementation. Vascular calcification will be measured at baseline and at 36 months of vitamin K supplementation by multi-slice CT scan. An additional EKG will be performed at 36 months of vitamin K supplementation to determine cardiac changes that may have occurred over the course of the study. Bilateral hand x-rays will be measured at 36 months of vitamin K supplementation, as will the administration of the Framingham OA questionnaire. Plasma 25-hydroxyvitamin D concentrations and urinary calcium and sodium will be measured at the same time points to be used as covariates in this assessment. In addition, 1,25-dihydroxyvitamin D will be measured at the beginning and end of the study. Other covariates collected throughout the study include age, weight, anthropometric data, physical activity, medication used, smoking, plasma lipids, insulin and measures of inflammation, B vitamins and dietary intakes. In addition, two tests of attention and concentration will be administered at 36 months of vitamin K supplementation. This trial will determine if supplemental vitamin K will reduce age-related bone loss, vascular calcification, osteoarthritis and concentration in elderly men and women, above that achieved by supplemental calcium and vitamin D alone.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory general population
* Dietary intake of vitamin K below 120 mcg

Exclusion Criteria:

* Unable to give informed consent
* Usual dietary intake of phylloquinone greater than 120 µg/d
* Usual dietary calcium intake greater than 1500 mg/d
* Usual dietary vitamin D intake greater than 1500 IU
* Women less than 5 years postmenopausal
* Femoral neck BMD (bone mineral density) at screening that is greater than 1.8 SD above or below an age-matched reference mean
* 24-hour calcium to creatinine ratio exceeding 300 mg/g for women or 350 mg/g for men
* Terminal illness
* Renal or liver disease requiring treatment
* Kidney stone in the past 5 years
* Current hyperparathyroidism
* Bilateral hip surgery
* Treatment with a bisphosphonate, calcitonin, estrogen progestin, androgen, tamoxifen, or fluoride (other than dental rinse), or any other treatment for osteoporosis in previous 3 months
* Warfarin or anticoagulant use in the past 12 months
* Nonambulation
* Known coronary disease, defined by myocardial infarction or unstable angina
* Prior open heart surgery
* Atrial fibrillation

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452
Dates: Start 2001-10; Study Completion 2006-10

PRIMARY OUTCOMES:
3 year change in bone mineral density at the hip
3 year change in coronary calcification score
Hand osteoarthritis score at final visit
Concentration and attention scores at final visit

SECONDARY OUTCOMES:
3 year change in biochemical measures of vitamin K status
3 year change in bone turnover
3 year change in measures of inflammation
Cardiac changes over 3 years
Difference in joint symptoms at final visit
3 year change in bone mineral density of the heel, spine and total body

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Booth, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Doherty TM, Asotra K, Fitzpatrick LA, Qiao JH, Wilkin DJ, Detrano RC, Dunstan CR, Shah PK, Rajavashisth TB. Calcification in atherosclerosis: bone biology and chronic inflammation at the arterial crossroads. Proc Natl Acad Sci U S A. 2003 Sep 30;100(20):11201-6. doi: 10.1073/pnas.1932554100. Epub 2003 Sep 19. PMID 14500910
- [Background] Jie KG, Bots ML, Vermeer C, Witteman JC, Grobbee DE. Vitamin K status and bone mass in women with and without aortic atherosclerosis: a population-based study. Calcif Tissue Int. 1996 Nov;59(5):352-6. doi: 10.1007/s002239900139. PMID 8849401
- [Background] Booth SL, Broe KE, Peterson JW, Cheng DM, Dawson-Hughes B, Gundberg CM, Cupples LA, Wilson PW, Kiel DP. Associations between vitamin K biochemical measures and bone mineral density in men and women. J Clin Endocrinol Metab. 2004 Oct;89(10):4904-9. doi: 10.1210/jc.2003-031673. PMID 15472183
- [Result] O'Donnell CJ, Shea MK, Price PA, Gagnon DR, Wilson PW, Larson MG, Kiel DP, Hoffmann U, Ferencik M, Clouse ME, Williamson MK, Cupples LA, Dawson-Hughes B, Booth SL. Matrix Gla protein is associated with risk factors for atherosclerosis but not with coronary artery calcification. Arterioscler Thromb Vasc Biol. 2006 Dec;26(12):2769-74. doi: 10.1161/01.ATV.0000245793.83158.06. Epub 2006 Sep 14. PMID 16973975
- [Derived] Shea MK, Booth SL, Miller ME, Burke GL, Chen H, Cushman M, Tracy RP, Kritchevsky SB. Association between circulating vitamin K1 and coronary calcium progression in community-dwelling adults: the Multi-Ethnic Study of Atherosclerosis. Am J Clin Nutr. 2013 Jul;98(1):197-208. doi: 10.3945/ajcn.112.056101. Epub 2013 May 29. PMID 23719555
- [Derived] Ma J, Ross AB, Shea MK, Bruce SJ, Jacques PF, Saltzman E, Lichtenstein AH, Booth SL, McKeown NM. Plasma alkylresorcinols, biomarkers of whole-grain intake, are related to lower BMI in older adults. J Nutr. 2012 Oct;142(10):1859-64. doi: 10.3945/jn.112.163253. Epub 2012 Sep 5. PMID 22955514
- [Derived] Shea MK, O'Donnell CJ, Vermeer C, Magdeleyns EJ, Crosier MD, Gundberg CM, Ordovas JM, Kritchevsky SB, Booth SL. Circulating uncarboxylated matrix gla protein is associated with vitamin K nutritional status, but not coronary artery calcium, in older adults. J Nutr. 2011 Aug;141(8):1529-34. doi: 10.3945/jn.111.139634. Epub 2011 May 31. PMID 21628633
- [Derived] Al Rajabi A, Peterson J, Choi SW, Suttie J, Barakat S, Booth SL. Measurement of menadione in urine by HPLC. J Chromatogr B Analyt Technol Biomed Life Sci. 2010 Sep 15;878(26):2457-60. doi: 10.1016/j.jchromb.2010.07.016. Epub 2010 Jul 29. PMID 20719580
- [Derived] Shea MK, Booth SL, Gundberg CM, Peterson JW, Waddell C, Dawson-Hughes B, Saltzman E. Adulthood obesity is positively associated with adipose tissue concentrations of vitamin K and inversely associated with circulating indicators of vitamin K status in men and women. J Nutr. 2010 May;140(5):1029-34. doi: 10.3945/jn.109.118380. Epub 2010 Mar 17. PMID 20237066
- [Derived] Shea MK, Gundberg CM, Meigs JB, Dallal GE, Saltzman E, Yoshida M, Jacques PF, Booth SL. Gamma-carboxylation of osteocalcin and insulin resistance in older men and women. Am J Clin Nutr. 2009 Nov;90(5):1230-5. doi: 10.3945/ajcn.2009.28151. Epub 2009 Sep 23. PMID 19776145
- [Derived] Shea MK, O'Donnell CJ, Hoffmann U, Dallal GE, Dawson-Hughes B, Ordovas JM, Price PA, Williamson MK, Booth SL. Vitamin K supplementation and progression of coronary artery calcium in older men and women. Am J Clin Nutr. 2009 Jun;89(6):1799-807. doi: 10.3945/ajcn.2008.27338. Epub 2009 Apr 22. PMID 19386744
- [Derived] Yoshida M, Jacques PF, Meigs JB, Saltzman E, Shea MK, Gundberg C, Dawson-Hughes B, Dallal G, Booth SL. Effect of vitamin K supplementation on insulin resistance in older men and women. Diabetes Care. 2008 Nov;31(11):2092-6. doi: 10.2337/dc08-1204. Epub 2008 Aug 12. PMID 18697901
- [Derived] Shea MK, Dallal GE, Dawson-Hughes B, Ordovas JM, O'Donnell CJ, Gundberg CM, Peterson JW, Booth SL. Vitamin K, circulating cytokines, and bone mineral density in older men and women. Am J Clin Nutr. 2008 Aug;88(2):356-63. doi: 10.1093/ajcn/88.2.356. PMID 18689371
- [Derived] Neogi T, Felson DT, Sarno R, Booth SL. Vitamin K in hand osteoarthritis: results from a randomised clinical trial. Ann Rheum Dis. 2008 Nov;67(11):1570-3. doi: 10.1136/ard.2008.094771. Epub 2008 Jul 14. PMID 18625626